CLINICAL TRIAL: NCT05632939
Title: A 1/2 Phase Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of ASKB589 in Combination With CAPOX and PD-1 Inhibitors in Patients With Advanced, and Unresectable Gastric/Esophagogastric Junction Cancer.
Brief Title: ASKB589 in Combination With CAPOX and PD-1 Inhibitors in Patients With Advanced, and Unresectable G/GEJ Cancer.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AskGene Pharma, Inc. (Industry)
Collaborators: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASK-LC-B589- Ib/II
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer; Gastroesophageal Cancer (GC)
Keywords: CLDN18.2; gastric cancer; gastroesophageal cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ASKB589 +CAPOX+Sintilimab/Tislelizumab (Experimental): Oxaliplatin: intravenous infusion, 130mg/m2, infusion for more than 3h, every 3 weeks for a cycle, infusion 6 cycles; Capecitabine: oral administration, 1000mg/m2, 2 times, 14 days, 7 days rest, every 3 weeks for a cycle; Sintilimab/Tislelizumab was administered intravenously at 200mg. The drug was administered once every 3 weeks, and the longest cumulative duration was 2 years.
  ASKB589 is administered intravenously at a fixed dose. the drug was given once every 3 weeks for a cycle, with the longest cumulative duration of 2 years.
  Interventions: Drug: ASKB589 +CAPOX+Sintilimab/Tislelizumab

INTERVENTIONS:
Drug: ASKB589 +CAPOX+Sintilimab/Tislelizumab — Oxaliplatin: intravenous infusion, 130mg/m2, infusion for more than 3h, every 3 weeks for a cycle, infusion 6 cycles; Capecitabine: oral administration, 1000mg/m2, 2 times, 14 days, 7 days rest, every 3 weeks for a cycle; Sintilimab/Tislelizumab was administered intravenously at 200mg. The drug was administered once every 3 weeks, and the longest cumulative duration was 2 years.
  ASKB589 is administered intravenously at a fixed dose. The drug was given once every 3 weeks for a cycle, with the longest cumulative duration of 2 years.

SUMMARY:
This was an open-label, phase 1/2 study to evaluate safety, tolerability, pharmacokinetics, and antitumor activity of ASKB589 in combination with CAPOX and PD-1 inhibitors in first-line treatment of patients with locally advanced, recurrent, or metastatic gastric and esophagogastric junction adenocarcinoma.

DETAILED DESCRIPTION:
A two-part, dose-escalation and expansion study of ASKB589 was initiated to determine the MTD, PK, PD, and efficacy in combination with chemotherapy and PD-1 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed unresectable locally advanced, recurrent, or metastatic adenocarcinoma of the gastric and gastroesophageal junction currently ineligible for surgery and radical radiotherapy.
2. Investigators determined that the present situation of the patient justifies chemotherapy plus immunotherapy as first-line treatment.
3. Tumor tissue samples are CLDN18.2 positive detected by central laboratory
4. ECOG performance status 0-1.
5. The results of the laboratory tests must meet all criteria
6. Life expectancy of at least 3 months.

Exclusion Criteria:

1. Known active central nervous system metastasis or suspected cancerous meningitis;
2. There are moderate to large amounts of abdominal and pleural fluid.
3. The presence of clinically uncontrollable third interspace fluid；
4. Patients with any other malignant tumors within the past 5 years.
5. Applicable to anti-HER-2 drug therapy；
6. Anti-CLDN18.2 antibody, anti-PD-1 antibody, or drug therapy at any time in the past；
7. Patients have received antitumor therapy during the first 4 weeks before study drug use;
8. Pregnant or lactating women; or women of childbearing age who have a positive blood pregnancy test during screening period; or women of childbearing age and their spouses who are unwilling to take effective contraceptive measures during the period of this clinical trial and within 6 months after the end of the clinical trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v5.0 | up to 21 days following last dose
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be presented.
The incidence and case number of DLT (Dose Limiting Toxicity) during observation period. | up to 21 days following last dose
  DLT is short for Dose Limiting Toxicity，dose-limiting describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Maximum Tolerated Dose (MTD） | up to 21 days following last dose
  The MTD was defined as the highest dose of ASKB589 not causing DLT in more than 33% of patients in the first treatment cycle.
The recommended dose | from date of treatment start until data cut-off, up to 2 years
  The recommended dose will be determined during the dose escalation and dose expansion stage of the study.

SECONDARY OUTCOMES:
Pharmacokinetics:maximum Plasma Concentration [Cmax] | Up to 21 days after injection
  Serum samples will be collected for Cmax analysis.
Pharmacokinetics:time to maximum observed plasma concentration (Tmax) | Up to 21 days after injection
  Serum samples will be collected for Tmax analysis.
Pharmacokinetics:elimination rate constant（Kel） | Up to 21 days after injection
  Serum samples will be collected for Kel analysis
Pharmacokinetics:terminal elimination half life (T1/2) | Up to 21 days after injection
  Serum samples will be collected for T1/2 analysis.
Pharmacokinetics:apparent volume of distribution (Vz/F) | Up to 21 days after injection
  Serum samples will be collected for Vz/F analysis.
Pharmacokinetics:Area Under Curve (AUC) | Up to 21 days after injection
  Serum samples will be collected for AUC analysis.
Pharmacokinetics: Mean ResidenceTime（MRT） | Up to 21 days after injection
  Serum samples will be collected for MRT analysis.
Pharmacokinetics: plasma clearance rate (CL) | Up to 21 days after injection
  Serum samples will be collected for CL analysis.
Pharmacokinetics: steady-state peak concentration (Css_max) | Up to 21 days after injection
  Serum samples will be collected for Css_max analysis.
Pharmacokinetics: time to steady-state peak concentration (Tss_max) | Up to 21 days after injection
  Serum samples will be collected for Tss_max analysis.
Pharmacokinetics: minimum value of steady plasma drug concentration（Css_min） | Up to 21 days after injection
  Serum samples will be collected for Css max analysis.
Evaluation of immunogenicity | from date of treatment start until data cut-off, up to 2 years
  Incidence of anti-drug antibodies (ADA)
Objective response rate（ORR） | from date of treatment start until disease progression,date of death or withdrawal from study,whichever came first, up to 2 years
  Evaluation of objective response rate assessed by RECIST 1.1
disease control rate（DCR) | from date of treatment start until disease progression,date of death or withdrawal from study,whichever came first, up to 2 years
  Evaluation of Disease control rate assessed by RECIST 1.1
Duration of Response（DOR） | from date of treatment start until disease progression,date of death or withdrawal from study,whichever came first, up to 2 years
  Duration of response assessed by RECIST 1.1
Progression free survival（PFS） | from date of treatment start until the date of disease progression or until death due to any causes, up to 2 years
  Progression of tumor will be measured by RECIST v1.1
Overall survival（OS） | from the date of treatment start until the documented date of death from any cause，up to 2 years.
  defined as the time from the date of treatment start until date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China